CLINICAL TRIAL: NCT01785433
Title: A Randomized, Open-Label, Repeat Dosing, Four-Period Crossover Study to Compare the Pharmacokinetics, Efficacy and Safety of Tiotropium Bromide Delivered Via Breath Actuated Inhaler (BAI), SPIRIVA® HandiHaler® and Respimat® Soft Mist™ Inhaler (SMI) in Subjects With COPD
Brief Title: To Compare the Pharmacokinetics of Tiotropium in Subjects With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: TBB-COPD-201
Record Dates: First submitted 2013-02-04; First posted 2013-02-07 (Estimated); Last update posted 2014-08-11 (Estimated); Status verified 2014-08

CONDITIONS: COPD
Keywords: COPD, pharmacokinetics, tiotropium
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Treatment ABCD (Experimental): The following treatments are to be studied in a 4-period, crossover design with once daily (QD) dosing for 7 days and at least 21 day washout period between treatments:
  Treatment A: Tiotropium HFA BAI 4.5 mcg/day
  Treatment B: Tiotropium HFA BAI 9.0 mcg/day
  Treatment C: SPIRIVA® HandiHaler® 18 mcg/day
  Treatment D: Spiriva® Respimat® 5 mcg/day
  Interventions: Drug: Tiotropium HFA BAI 4.5 mcg; Drug: Tiotropium HFA BAI 9.0 mcg; Drug: SPIRIVA® HandiHaler® 18 mcg/day; Drug: Spiriva® Respimat® 5 mcg/day
- Treatment BDAC (Experimental): The following treatments are to be studied in a 4-period, crossover design with once daily (QD) dosing for 7 days and at least 21 day washout period between treatments:
  Treatment B: Tiotropium HFA BAI 9.0 mcg/day
  Treatment D: Spiriva® Respimat® 5 mcg/day
  Treatment A: Tiotropium HFA BAI 4.5 mcg/day
  Treatment C: SPIRIVA® HandiHaler® 18 mcg/day
  Interventions: Drug: Tiotropium HFA BAI 4.5 mcg; Drug: Tiotropium HFA BAI 9.0 mcg; Drug: SPIRIVA® HandiHaler® 18 mcg/day; Drug: Spiriva® Respimat® 5 mcg/day
- Treatment CADB (Experimental): The following treatments are to be studied in a 4-period, crossover design with once daily (QD) dosing for 7 days and at least 21 day washout period between treatments:
  Treatment C: SPIRIVA® HandiHaler® 18 mcg/day
  Treatment A: Tiotropium HFA BAI 4.5 mcg/day
  Treatment D: Spiriva® Respimat® 5 mcg/day
  Treatment B: Tiotropium HFA BAI 9.0 mcg/day
  Interventions: Drug: Tiotropium HFA BAI 4.5 mcg; Drug: Tiotropium HFA BAI 9.0 mcg; Drug: SPIRIVA® HandiHaler® 18 mcg/day; Drug: Spiriva® Respimat® 5 mcg/day
- Treatment DCBA (Experimental): The following treatments are to be studied in a 4-period, crossover design with once daily (QD) dosing for 7 days and at least 21 day washout period between treatments:
  Treatment D: Spiriva® Respimat® 5 mcg/day
  Treatment C: SPIRIVA® HandiHaler® 18 mcg/day
  Treatment B: Tiotropium HFA BAI 9.0 mcg/day
  Treatment A: Tiotropium HFA BAI 4.5 mcg/day
  Interventions: Drug: Tiotropium HFA BAI 4.5 mcg; Drug: Tiotropium HFA BAI 9.0 mcg; Drug: SPIRIVA® HandiHaler® 18 mcg/day; Drug: Spiriva® Respimat® 5 mcg/day

INTERVENTIONS:
Drug: Tiotropium HFA BAI 4.5 mcg
Drug: Tiotropium HFA BAI 9.0 mcg
Drug: SPIRIVA® HandiHaler® 18 mcg/day
Drug: Spiriva® Respimat® 5 mcg/day

SUMMARY:
The primary objective of this study is to assess and compare the pharmacokinetics (PK) of Tiotropium delivered via Breath Actuated Inhaler (BAI) (4.5 mcg/day or 9.0 mcg/day), SPIRIVA®, HandiHaler®, (18 mcg/day) and Respimat® Soft Mist™ Inhaler (SMI) (5.0 mcg/day) following repeat dosing for 7 days in subjects with COPD.

DETAILED DESCRIPTION:
This multicenter study consists of a Screening Visit (3 to 14 days prior to randomization); 4 multiple-dose (7-day) Treatment Periods, each consisting of a 2-night/3-day inpatient stay (Day 6 to Day 8); and a Final Visit. A washout period of at least 21 days will occur between each Treatment Period. The Final/ Early Termination Visit will occur 6-8 days following the last Treatment Period or upon early discharge from the study.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent signed and dated by the subject before conducting any study related procedure
2. Male or female subjects 40 -80 years of age, as of the Screening Visit
3. Diagnosis of COPD as defined by the GOLD (Global Initiative for Chronic Obstructive Lung Disease) Guidelines
4. A pre-bronchodilator Peak Inspiratory Flow (PIF) rate≥ 30 L/ min as measured with the In-Check™ DIAL training device.
5. A measured post-bronchodilator (ipratropium bromide) forced expiratory volume in one second (FEV1) >30% and <80% of predicted normal for height, age and gender at the Screening Visit (SV). Third National Health and Nutrition Examination Survey 1988-1994 (NHANES III) predicted values will be used and adjustments to predicted values will be made for African-American subjects.
6. A measured post-bronchodilator (ipratropium bromide) FEV1/Forced Vital Capacity (FVC) <0.70 at the Screening Visit (SV)
7. If female, is currently not pregnant, breast feeding, or attempting to become pregnant (for 4 weeks before the Screening Visit (SV) and throughout the duration of the study), and is of

   * Non-childbearing potential, defined as:

     * ≥1 year post-menopausal or
     * Surgically sterile (tubal ligation, bilateral oophorectomy, salpingectomy, or hysterectomy) or is of
   * Childbearing potential, has a negative serum pregnancy test, and is willing to commit to using a consistent and acceptable method of birth control as defined below for the duration of the study:

     * Systemic contraception used for ≥1 month prior to screening, including birth control pills, transdermal patch, vaginal ring, implants, or injectables or
     * Double barrier methods (condoms, cervical cap, diaphragm, and vaginal contraceptive film with spermicide) or
     * Intrauterine device (IUD) with a low failure rate defined as <1% per year (use of copper IUDs are excluded) or is of

       * Childbearing potential and not sexually active, has a negative serum pregnancy test, and is willing to commit to using a consistent and acceptable method of birth control as defined above for the duration of the study, in the event the subject becomes sexually active
8. Current or ex-smoker with ≥10 pack-year smoking history
9. Subject is free of any concomitant conditions or treatment that could interfere with study conduct, influence the interpretation of study observations/results, or put the subject at increased risk during the study
10. Able to perform technically acceptable and reproducible spirometry per study guidelines as defined in the protocol and study procedures manual.
11. Able to demonstrate the proper inhalation techniques required for correct use of all delivery devices required in the study
12. Capable of understanding the requirements, risks, and benefits of study participation, and, as judged by the investigator, capable of giving informed consent and being compliant with all study requirements

Exclusion Criteria:

1. Pregnancy, nursing, or plans to become pregnant or donate gametes (ova or sperm) for in vitro fertilization during the study period or for 30 days following the subject's last study related visit (for eligible subjects only, if applicable).
2. History or current evidence (as determined by medical history, physical examination, clinical laboratory assessments and ECG) of a clinically significant or uncontrolled disease including, but not limited to: cardiovascular (e.g., uncontrolled hypertension, congestive heart failure, known aortic aneurysm, clinically significant cardiac arrhythmia or coronary heart disease), hepatic, renal, haematological, neuropsychological, endocrine (e.g., uncontrolled diabetes mellitus, uncontrolled thyroid disorder, Addison's disease, Cushing's syndrome), gastrointestinal (e.g., poorly controlled peptic ulcer, gastroesophageal reflux disease) or pulmonary (other than COPD such as asthma, sarcoidosis, non-cystic fibrosis (CF) bronchiectasis, cystic fibrosis, bronchopulmonary dysplasia or a diagnosis of alpha 1-antitrypsin deficiency). Significant is defined as any disease that, in the opinion of the investigator, would put the safety of the subject at risk through participation, or which could affect the endpoint analysis if the disease/condition exacerbated during the study.
3. History of and/or current diagnosis of asthma
4. History of a life-threatening COPD exacerbation - defined for this protocol as a COPD episode that required intubation and/or was associated with hypercapnia, respiratory arrest or hypoxic seizures
5. Thoracotomy with pulmonary resection
6. Current congestive heart failure, history or current evidence of myocardial infarction (within 3 yrs of the Screening Visit [SV]), or history or current evidence of ischemic heart disease, including a diagnosis on screening ECG.
7. History or current evidence of clinically significant cardiac arrhythmia, including a diagnosis on screening ECG.
8. Presence of angle-closure glaucoma
9. History of malignancy (excluding basal cell carcinoma) within the past 5 years, regardless of the clinical significance or current stability of the disease
10. Known history or any current evidence of renal impairment or urinary retention (e.g., bladder outlet obstruction). This includes abnormal renal function test results at screening.
11. Presence of symptomatic prostatic hyperplasia
12. History of silent infections, including positive tests for human immunodeficiency virus 1, human immunodeficiency virus 2, Hepatitis B, Hepatitis C, or tuberculosis.
13. Occurrence of any upper or lower respiratory infection, including but not limited to the common cold and flu, sinusitis,tonsillitis, pneumonia, bronchitis, or an ear infection (including otitis media and externa) which is not resolved by 14 days prior to randomization
14. Occurrence of a COPD exacerbation which is not resolved by 14 days prior to randomization i. Note: An exacerbation of COPD is defined as any worsening of the subject's baseline COPD symptoms requiring any treatment other than rescue albuterol/salbutamol/ipratropium or the subject's regular maintenance treatment. This includes requiring the use of systemic corticosteroids and/or emergency room visit or hospitalization, a change in subject's regular, or the addition of other medications used to treat COPD symptoms.
15. Subjects who require oxygen therapy and in the investigator's opinion, will be unable to abstain from the use of oxygen therapy during testing
16. Subjects who have started or stopped an exercise rehabilitation program within 4 weeks of the Screening Visit (SV)
17. Known or suspected hypersensitivity or idiosyncratic reaction to tiotropium, or to any ingredients used in the study medication formulations
18. Severe allergy to milk protein
19. Significant adverse drug reactions, including allergy or hypersensitivity reactions, to atropine or any anticholinergic substance related pharmacologically to atropine (e.g., ipratropium or oxitropium)
20. Use of any prohibited concomitant medications within the prescribed (per protocol) withdrawal periods prior to the Screening Visit
21. Treatment with orally administered (excluding orally inhaled) β-adrenergics (i.e., oral salbutamol)
22. Treatment with β-adrenergic receptor antagonists (e.g. non-selective β-receptor blocking agents like β-blocking anti-hypertensive products) administered by any route. The single exception is that cardioselective β1-adrenergic receptor antagonists (e.g. atenolol, metoprolol, bisoprolol) are permitted provided that subjects have been on a stable dose for at least 1 week prior to the screening visit and subjects are expected to be able to maintain the same dose throughout the study.
23. Treatment with drugs commonly recognized to prolong the QTc interval (e.g., quinolones, amiodarone, disopyramide, quinidine, sotalol, chlorpromazine, haloperidol, ketoconazole, terfenadine, cisapride and terodiline)
24. Treatment with any known cytochrome P450 (CYP) 2D6 or cytochrome P450 (CYP) 3A4 inhibitors (e.g., quinidine, ketoconazole and gestodene) within 30 days prior to the Screening Visit (SV)
25. Initiation or change in dose of inhaled corticosteroids within the last 6 weeks prior to the Screening Visit (SV), and /or not expected to maintain a stable dose of inhaled corticosteroids during the course of the study.
26. Initiation or change in dose of oral or systemic corticosteroids within the last 6 weeks prior to the Screening Visit (SV) , unable to maintain a stable dose of oral or systemic corticosteroids during the course of the study, or a dose of oral or systemic corticosteroids in excess of the equivalent of 10 mg of prednisone per day. [Note that oral steroid bursts completed 6 weeks or more prior to screening are acceptable.]
27. Exposure to any investigational drug within 30 days or six half-lives (whichever is greater) prior to the Screening Visit (SV)
28. Plans to donate or has donated plasma or blood within 1 month prior to the Screening Visit (SV). This does not include small blood volumes taken for diagnostic purposes. Plans to donate plasma or blood within 3 months following study completion
29. Has a history of alcohol and/or substance abuse within the past 5 years
30. Vulnerable subjects (e.g., persons kept in detention)
31. The subject is an employee of the study site or has an immediate family member or household member involved with the conduct of the study (including participation in the study).

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2013-01; Primary Completion 2013-07 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration-time curve (AUC0-24h) | From time 0 to 24 hours on Day 7
  To evaluate the PK of Tiotropium Hydrofluoroalkane (HFA) Breath Actuated Inhaler (BAI) (4.5 mcg/day and 9 mcg/day) to SPIRIVA® HandiHaler® and Spiriva® Respimat®
Maximum observed plasma concentration (Cmax) | From time 0 to 24 hours on Day 7
  To evaluate the PK of Tiotropium HFA BAI (4.5 mcg/day and 9 mcg/day) to SPIRIVA® HandiHaler® and Spiriva® Respimat®

SECONDARY OUTCOMES:
Area under the plasma concentration-time curve (AUC 0-t) | From time 0 to the time of the last quantifiable concentration as measured up to 24 hrs on Day 7
  To evaluate the PK of Tiotropium HFA BAI (4.5 mcg/day and 9 mcg/day) to SPIRIVA® HandiHaler® and Spiriva® Respimat®
Time at which the maximum plasma concentration was observed (tmax) | From time 0 to 24 hours on Day 7
  To evaluate the PK of Tiotropium HFA BAI (4.5 mcg/day and 9 mcg/day) to SPIRIVA® HandiHaler® and Spiriva® Respimat®
Occurrence of Adverse Events | From signing of the Informed Consent Form until the final visit (approximately 6 to 8 days following the last treatment period)
  The adverse event frequency, intensity, severity and relationship to the study drug will be recorded.

CONTACTS AND LOCATIONS:
Locations (5):
- Germany (5):
  - Teva Investigational Site 32170, Berlin
  - Teva Investigational Site 32169, Gauting
  - Teva Investigational Site 32171, Großhansdorf
  - Teva Investigational Site 32167, Mannheim
  - Teva Investigational Site 32168, Wiesbaden